CLINICAL TRIAL: NCT01526343
Title: A Comparison of Traditional Arrhythmia Assessment With the Use of Continuous Monitoring to Quantify Postoperative Arrhythmia Burden Following Surgical Treatment of Atrial Fibrillation- Medtronic Reveal XT Study
Brief Title: Medtronic Reveal XT Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Jennifer Bell, Manager of Research, Cardiothoracic Surgery, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201105015
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
Keywords: Patients
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reveal XT (Experimental)
  Interventions: Device: Reveal XT implantation

INTERVENTIONS:
Device: Reveal XT implantation — The implantation of the Reveal XT device will be performed at the time of surgery before the planned median sternotomy or thoracotomy.

SUMMARY:
While surgical treatment for atrial fibrillation (AF) has been performed for over 20 years, virtually all of the historical series reported only the recurrence of symptomatic AF and have used only intermittent electrocardiogram (ECG) follow-up. This study compares the use of traditional arrhythmia assessment (ECG and 24-hour holter monitoring) with the use of the Medtronic Reveal XT device to continuously record heart rhythm to quantify postoperative arrhythmia burden following surgical treatment for AF in patients undergoing either lone or concomitant heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing planned, elective AF surgery, either as a stand-alone procedure or as a concomitant cardiac operation.
2. Patients will have either a Cox-Maze procedure (full-biatrial lesion set) or surgical pulmonary vein isolation (PVI).
3. Patients 18 years or older.
4. All eligible patients will be considered, regardless of gender or race.
5. Patients able and willing to provide informed consent and willing to comply with the required interval follow-up.

Exclusion Criteria:

1. Patients with a preoperative permanent pacemaker.
2. Patients with a projected lifespan of less than six months.
3. Patients requiring emergent cardiac surgery.
4. Patients unwilling or unable to give written informed consent.
5. Patients undergoing a right atrial or left atrial lesion set procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J Damiano, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 47 consecutive patients who received an implantable loop recorder (ILR) after a surgical ablation procedure were followed between August 2011 and January 2014. Patients with AF who were scheduled to undergo elective surgical ablation procedure that included a CM IV lesion set or pulmonary vein isolation were eligible.
Period: Overall Study
Arm/Group | Reveal XT
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reveal XT
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of ATA (Atrial Tachyarrhythmias) Episodes and Burden, Determined at Defined Postoperative Intervals
Time Frame: ILR monitoring obtained at 3, 6 and 12 months
Measure: Number; unit: ATA episodes
Arm/Group | Reveal XT
Number analyzed (Participants) | 47
ATA episodes
  Count of total ATAs | 20,878
  Count of reviewed and confirmed ATAs | 1,034

2. Primary Outcome: Freedom From Atrial Tachyarrhythmias (ATAs)
Time Frame: ILR monitoring at 12 months
Population: Participants with available data at 1 year and who were compliant with use of each device.
Measure: Number; unit: Participants
Arm/Group | Reveal XT
Number analyzed (Participants) | 46
Participants
  Freedom from ATAs at 1 year, ILR device: number analyzed (Participants) | 42
  Freedom from ATAs at 1 year, ILR device | 37
  Freedom from ATAs at 1 year, Holter monitor: number analyzed (Participants) | 35
  Freedom from ATAs at 1 year, Holter monitor | 33
  Freedom from ATAs at 1 year, ECG: number analyzed (Participants) | 39
  Freedom from ATAs at 1 year, ECG | 37

ADVERSE EVENTS:
Groups:
- Reveal XT: Reveal XT implantation: The implantation of the Reveal XT device will be performed at the time of surgery before the planned median sternotomy or thoracotomy.
  No reportable adverse events occurred.
Arm/Group | Reveal XT
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No